CLINICAL TRIAL: NCT05813470
Title: A Phase III, Randomized, Multicenter, Double-blind, Two-armed, Parallel, Active-controlled, Equivalency Clinical Trial to Compare Efficacy and Safety of Omalizumab (CinnaGen, Iran) in Comparison to Xolair® (Genentech, Inc., USA And Novartis Pharmaceuticals Corp, Switzerland) in Patients With Uncontrolled Moderate to Severe Allergic Asthma
Brief Title: Efficacy and Safety of Zerafil® (Omalizumab) in Participants With Uncontrolled Moderate to Severe Allergic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMA.CIN.EI.97.III
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Allergic Asthma; Uncontrolled Moderate to Severe
Keywords: Asthma; Omalizumab; Exacerbation Rate; Monoclonal
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omalizumab (CinnaGen) (Experimental): Omalizumab (CinnaGen) was administered every 2 or 4 weeks to provide a dose of at least 0.016 mg/kg/IgE for a duration of 28 weeks
  Interventions: Biological: Omalizumab (CinnaGen)
- Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland) (Active Comparator): Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland) was administered every 2 or 4 weeks to provide a dose of at least 0.016 mg/kg/IgE for a duration of 28 weeks
  Interventions: Biological: Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland)

INTERVENTIONS:
Biological: Omalizumab (CinnaGen) — Omalizumab (CinnaGen, Iran) was administered via subcutaneous injection
  Other Names: Zerafil®
  Arms: Omalizumab (CinnaGen)
Biological: Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland) — Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland) was administered via subcutaneous injection
  Other Names: Xolair®
  Arms: Omalizumab (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Omalizumab produced by CinnaGen compared with Xolair® (Genentech, Inc., USA And Novartis Pharmaceuticals Corp, Switzerland) in subjects with uncontrolled Moderate to Severe Allergic Asthma

All the participants will receive one of the following regimens:

Omalizumab (CinnaGen) or Xolair® (Genentech, Inc., USA And Novartis Pharmaceuticals Corp, Switzerland), as subcutaneous injections, Omalizumab was administered every 2 or 4 weeks to provide a dose of at least 0.016 mg/kg/IgE for a duration of 28 weeks

The primary objective of this study is to assess whether the efficacy of Omalizumab (CinnaGen, Iran) is equivalent to Xolair® (Genentech, Inc., USA and Novartis Pharmaceuticals Corp, Switzerland) as measured by rate of protocol-defined asthma exacerbations during the 28-week treatment period

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent and to be compliant with the schedule of protocol assessments
2. Positive skin prick or in vitro reactivity test to ≥ 1 perennial aeroallergen
3. Total serum IgE level of ≥30 to ≤700 IU/ml.
4. Moderate to Severe persistent asthma requiring regular treatment with high dose of inhaled corticosteroid (ICS) (GINA 2019 step 4 treatment).
5. Body weight of ≥30 to ≤150
6. History of one of these 2 items during the past 12 months:

   * At least 2 asthma exacerbations which needed systemic corticosteroids, (≥30 days prior to screening)
   * Severe asthma exacerbation in which peak expiratory flow (PEF) or FEV1 was less than 60% of the patient best result and needed systemic corticosteroids and hospitalization or emergency department visit, (≥30 days prior to screening)

Exclusion Criteria:

1. Smoking history of ≥10 pack-years
2. Chronic use of corticosteroids (use of 20 to 30 mg prednisolone for more than 3 weeks) or other immunosuppressant due to other disease except asthma such as autoimmune or collagen vascular disease and etc.
3. Treatment with omalizumab in the 12 months before screening
4. History of severe allergic or anaphylactic reactions to Omalizumab
5. Active lung disease other than asthma
6. Acute upper respiratory tract infection within 1 month before screening
7. Unable to perform spirometry test and other tests needed in the trial
8. Female subjects who are not willing to practice effective contraception (as defined by the investigator) during the study
9. Nursing mothers, pregnant women, and women who planned to become pregnant while on study
10. Participation in any other investigational study within 6 months prior to randomization
11. Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that was likely to affect the subject's ability to comply with the study protocol
12. Persons have an asthma exacerbation requiring intubation in the 12 months before screening
13. Unexpected events that prevent patient entering the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of protocol-defined asthma exacerbations during the 28-week treatment period | 28 weeks
  Protocol-defined asthma exacerbation (PDAE) is defined as worsening asthma symptoms requiring treatment with 40-50 mg oral corticosteroids for 3-7 days; for patients receiving long-term Oral Corticosteroids, an exacerbation is a 20-mg or more increase in the average daily dose of oral prednisolone (or a comparable dose of another oral corticosteroids)

SECONDARY OUTCOMES:
Change in Asthma Control Test (ACT) score from baseline to the end (last four weeks) over the 28 weeks | 28 weeks
  Asthma Control Test (ACT) scores range from 5-25 (higher is better). Scores of 20-25 are classified as well-controlled asthma; 16-19 as not well-controlled; and 5-15 as very poorly controlled asthma.
Change in spirometry measures (FEV1) in 28 weeks | 28 weeks
  FEV1: Forced Expiratory Volume in the first second of exhalation
Immunogenicity Assessment | 28 weeks
  Number of participants positive for anti-drug antibodies at weeks 16 and 28
Evaluation of adverse events during 28 weeks | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Esmaeil Idani, Pulmonologist, Principal Investigator — NRITLD, Shahid Beheshti University of Medical Sciences
Locations (22):
- Iran (22):
  - Golestan Hospital, Ahvāz
  - Imam Khomeini, Ahvāz
  - Khorshid Hospital, Isfahan
  - Dr.Tavakoul Office, Karaj
  - Afzaalipour Hospital, Kerman
  - Dr.Mirsadraei Office, Mashhad
  - Qaem Hospital, Mashhad
  - Dr.Qalebaqi Office, Rasht
  - Razi Hospital, Rasht
  - Imam Khomeini Hospital, Sari
  - Imam Reza Hospital, Shiraz
  - Imam Reza Hospital, Tabriz
  - Baqiatallah Hospital, Tehran
  - Firouzgar Hospital, Tehran
  - Imam Khomeini Hospital, Tehran
  - Jihad Academic Asthma and Allergy Clinic, Tehran
  - Masih Hospital, Tehran
  - Modares Hospital, Tehran
  - Rasoul Akram Hospital, Tehran
  - Shariati Hospital, Tehran
  - Sadoghi Hospital, Yazd
  - Valiasr Hospital, Zanjān

REFERENCES:
- [Derived] Ghanei M, Ghalebaghi B, Sami R, Torabizadeh M, Mirsadraee M, Amra B, Tavakol M, Raji H, Fallahpour M, Kiani A, Abedini A, Jabbari Azad F, Mahdaviani SA, Attaran D, Samet M, Tavana S, Haddadzadeh Shoushtari M, Nazari J, AghaeiMeybodi F, Fazlollahi MR, Ghasemi R, Sabzvari A, Kafi H, Idani E. Efficacy and safety of a proposed omalizumab biosimilar compared to the reference product in the management of uncontrolled moderate-to-severe allergic asthma: a multicenter, phase III, randomized, double-blind, equivalency clinical trial. Front Immunol. 2024 Jul 29;15:1425906. doi: 10.3389/fimmu.2024.1425906. eCollection 2024. PMID 39136011